CLINICAL TRIAL: NCT06688175
Title: Intensity-modulated Radiotherapy Combined With Lobaplatin-based Concurrent Chemotherapy in the Treatment of Elderly Patients With Nasopharyngeal Carcinoma
Brief Title: IMRT Combined With Lobaplatin-based CCRT in Nasopharyngeal Carcinoma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, San-Gang Wu, Clinical Professor, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY062
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Neoplasms; Elderly; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): in the treatment of elderly patients with nasopharyngeal carcinoma
  Interventions: Drug: IMRT combined with lobaplatin-based concurrent chemotherapy

INTERVENTIONS:
Drug: IMRT combined with lobaplatin-based concurrent chemotherapy — IMRT combined with two cycles of lobaplatin-based concurrent chemotherapy

SUMMARY:
This prospective, multicenter, single-arm, open-label phase II clinical study aimed to investigate the efficacy and safety of intensity-modulated radiotherapy combined with lobaplatin-based concurrent chemotherapy in the treatment of elderly patients with nasopharyngeal carcinoma

DETAILED DESCRIPTION:
Lobaplatin, as a third-generation platinum-based chemotherapeutic agent, demonstrates equivalent therapeutic efficacy to cisplatin but significantly lower toxicity. Preliminary clinical trials have confirmed that lobaplatin shows substantial effectiveness in treating various cancers including breast cancer, esophageal cancer, colorectal cancer, and cervical cancer. Importantly, lobaplatin does not exhibit cross-resistance with cisplatin or carboplatin, indicating a promising application prospect.

Currently, lobaplatin has demonstrated clear efficacy in non-elderly nasopharyngeal carcinoma (NPC) chemotherapy. Guo Xiang et al. have confirmed that for non-elderly NPC patients, induction chemotherapy with lobaplatin followed by concurrent chemoradiotherapy may be a treatment option for locally advanced NPC. However, there is very limited research reporting on the use of lobaplatin in elderly NPC patients.

Based on the above theoretical considerations and our research results, lobaplatin shows good safety and reliable efficacy in treating elderly NPC, with minimal gastrointestinal reactions and low incidence of renal, neurotoxic, and ototoxic effects. This approach significantly enhances the quality of life for locally advanced elderly NPC patients. Therefore, the efficacy and safety of lobaplatin in concurrent chemotherapy for elderly NPC deserve further investigation. This study aims to evaluate the recent efficacy, safety, and toxic side effects of lobaplatin combined with intensity-modulated radiotherapy in the treatment of elderly NPC. Designed as a multicenter, open-label, prospective study, it aims to verify whether lobaplatin is an effective concurrent chemotherapeutic agent for elderly NPC, while further improving the quality of life for these patients under guarantees of therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed differentiated non-keratinizing carcinoma and undifferentiated non-keratinizing carcinoma;
* Stage II-IVa (UICC 8th edition);
* Acceptable induction chemotherapy and Tarceva targeted therapy;
* No history of other malignant tumors;
* Male or female, aged 65-80 years.
* Liver function: Total bilirubin ≤ Upper Limit of Normal (ULN); AST and ALT ≤ 2.5 times ULN; Alkaline phosphatase ≤ 5 times ULN;
* Renal function: Creatinine clearance ≥ 60 ml/min or Creatinine ≤ 1.5 × ULN;
* Hematological tests: Absolute Neutrophil Count (ANC) ≥ 2 × 10^9/L, Platelet count ≥ 100 × 10^9/L, and Hemoglobin ≥ 9 g/dL;
* No severe dysfunction of vital organs such as heart and lung;
* PS score ≤ 2 points

Exclusion Criteria:

* Distant metastases detected before treatment;
* Refusal to sign the informed consent form;
* Patients who cannot comply with regular follow-up due to psychological, social, family, or geographical reasons;
* Simultaneously receiving other experimental treatments in clinical trials (during the treatment phase of clinical research);
* Severe, uncontrolled infections or medical conditions;
* Vital organ dysfunction, decompensated heart, lung, kidney, or liver failure, unable to tolerate radiotherapy and chemotherapy;
* Laboratory tests: Total bilirubin > Upper Limit of Normal (ULN); AST and/or ALT > 1.5 times ULN with alkaline phosphatase > 2.5 times ULN;
* Factors affecting drug administration, distribution, metabolism, and excretion, such as mental abnormalities, central nervous system abnormalities, chronic diarrhea, ascites, pleural effusion, etc.;
* Long-term use of immunosuppressants after organ transplantation;
* Patients with a history of other malignant tumors before enrollment.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 months
  ORR encompasses both CR and PR.

SECONDARY OUTCOMES:
Safety | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Overall survival (OS) | 3 years
  OS was defined as the time of NPC diagnosis until death from any cause.
Locoregional relapse-free survival (LRFS) | 3 years
  LRFS was measured as the duration time from the diagnosis of nasopharyngeal carcinoma to the occurrence of relapse in the nasopharynx or neck lymph nodes or until the last follow-up.
Distant metastasis-free survival (DMFS) | 3 years
  DMFS was defined as the duration time of nasopharyngeal carcinoma diagnosis to the time of distant metastasis or the last follow-up.
Progression-free survival (PFS) | 3 years
  PFS was referred to as the time from nasopharyngeal carcinoma diagnosis to the date of disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No